CLINICAL TRIAL: NCT01052688
Title: Noninvasive Screening for Fetal Chromosomal Aneuploidy and Abnormality: Assay Development & Optimization in Affected Pregnancies
Brief Title: Noninvasive Screening for Affected Pregnancies: Assay Development & Optimization in Affected Pregnancies
Acronym: CHARMM-AP
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM T21-305
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2020-04

CONDITIONS: Down Syndrome; Aneuploidy
Keywords: Down syndrome, aneuploidy, amniocentesis, chorionic villus sampling, Trisomy
MeSH Terms: conditions — Down Syndrome; Aneuploidy; Trisomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, white blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant Women: Pregnant women who have been definitively diagnosed as carrying a fetus with aneuploidy.
  Interventions: Other: Maternal blood draw of 30 to 50ml

INTERVENTIONS:
Other: Maternal blood draw of 30 to 50ml — Maternal blood draw of 30 to 50mls during pregnancy. Blood may be drawn up to 5 times during the pregnancy between weeks 8 and 36 gestation.

SUMMARY:
To collect samples for the purpose of developing and optimizing an in vitro noninvasive prenatal diagnostic (NIPD) test. The NIPD test employs circulating cell free (ccff) DNA extracted from whole blood samples collected from women who are pregnant with a fetus previously determined to have a chromosomal abnormality. The NIPD result will be compared to the standard test results obtained from other test methods such as karyotype, FISH, QF-PCR, and/or any commercially available NIPD test.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female
* Subject is 18 years or older
* Subject is no less than 8 and no more than 36 weeks gestation
* Subject provides a signed and dated informed consent
* Subject agrees to provide one or more 30-50mL blood sample(s) in accordance with the protocol
* Subject has a current pregnancy in which the fetus is known to have chromosomal aneuploidy (e.g. T13, T18, T21)

Exclusion Criteria:

* Non-singleton pregnancy in which only one fetus is known to have a chromosomal aneuploidy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who have been definitively diagnosed by amniocentesis, CVS or QF/PCR as carrying a fetus with aneuploidy
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-11; Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
NIPD result compared to standard test results | baseline
  Result of NIPD test will be compared to the standard test results obtained by karyotype, FISH, QF-PCR, and/or commerical NIPD result.

CONTACTS AND LOCATIONS:
Overall Officials: Juan-Sebastian Saldivar, M.D., Study Director — Sequenom, Inc.
Locations (10):
- United States (10):
  - Perinatal Care Associates, Phoenix, Arizona
  - St. Joseph's Hospital and medical Center, Phoenix, Arizona
  - Sharp Grossmount, San Diego, California
  - IGO, San Diego, California
  - San Diego Perinatal Center, San Diego, California
  - Women's Healthcare at Frost Street, San Diego, California
  - Reiter, Hill, Johnson and Nevin, Washington D.C., District of Columbia
  - Fetal Diagnostic Institute of the Pacific, Honolulu, Hawaii
  - Spectrum Health, Grand Rapids, Michigan
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
Samples and data are used in research and development of a noninvasive prenatal test. However, sample data used in publications will be shared as per requirements of the journal.